CLINICAL TRIAL: NCT06886971
Title: Strategies to AchieVe Viral Suppression for Youth With HIV (The SAVVY Study)
Brief Title: Strategies to AchieVe Viral Suppression for Youth With HIV
Acronym: SAVVY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00421059; R01MH134724 (NIH)
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Human Immunodeficiency Virus (HIV) Infection
Keywords: adolescents; long-acting antiretroviral treatment; youth; young adu;ts; viral suppression; effectiveness
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The SAVVY intervention includes CHOICE counseling and shared decision-making regarding ART preference (informed by the evidence-based HIV-ASSIST) and facilitating long-acting injectable ART (LAI-ART) access to that choice through the deployment of the SLAT team. HIV-ASSIST is an interactive tool that offers clinicians comprehensive, individualized validated patient-specific antiretroviral (ARV) decision support along with evidence-based supporting educational material. The free online, interactive tool is designed to augment interpretation of current HIV clinical practice guidelines (CPG). SAVVY will use HIV-ASSIST and CHOICE counseling (an evidence-based strategy addressing patient knowledge about effectiveness, advantages, and identified needs) to facilitate selection of participants preferred treatment strategy and then evaluate outcomes (HIV (viral suppression) and quality of life indicators)). SAVVY will also evaluate uptake of long-acting injectable over the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virally suppressed at entry (VL<50 copies/mL) (Other): Participants are on ART and are currently virally suppressed. Participants will undergo CHOICE counseling and determine if the participant prefers to stay on oral ART or switch to LAI-ART. The SAVVY long-acting access team (SLAT) will facilitate prior authorizations and other logistic matters needed to access LAI-ART. The study will not provide drug.
  Participants will participate in a baseline, 3, 6, 9 and 12 month detailed assessment of viral suppression and quality of life indicators, etc.
  Interventions: Other: The SAVVY intervention includes CHOICE counseling and shared decision-making regarding ART preference (informed by the evidence-based HIV-ASSIST) and facilitating LA-ART access
- Not virally suppressed at entry (VL >= 50 copies/mL) (Other): Participants are on ART and are currently not virally suppressed. The participants will undergo CHOICE counseling and determine if the participant prefers to stay on oral ART or switch to LAI-ART. As the participant will not be able to switch to LAI-ART given the viremic state, the participant will have q2 week monitoring (for 3 months) of the viral load and if the participant becomes suppressed will then be offered CHOICE counseling again and can select at that point if the participant wants to stay on oral or transition to LAI-ART. The SAVVY long-acting access team will facilitate prior authorizations and other logistic matters needed to access LAI-ART. The study will not provide drug.
  If the participant has not become suppressed by 3 months the participant would continue to be monitored by standard of care practices.
  Participants will participate in a baseline, 3, 6, 9 and 12 month detailed assessment of viral suppression and quality of life indicators, etc.
  Interventions: Other: The SAVVY intervention includes CHOICE counseling and shared decision-making regarding ART preference (informed by the evidence-based HIV-ASSIST) and facilitating LA-ART access

INTERVENTIONS:
Other: The SAVVY intervention includes CHOICE counseling and shared decision-making regarding ART preference (informed by the evidence-based HIV-ASSIST) and facilitating LA-ART access — The SAVVY intervention includes CHOICE counseling and shared decision-making regarding ART preference (informed by the evidence-based HIV-ASSIST) and facilitating LA-ART access to that choice through the deployment of the SLAT team. HIV-ASSIST is an interactive tool that offers clinicians comprehensive, individualized validated patient-specific ARV decision support along with evidence-based supporting educational material. The free online, interactive tool is designed to augment interpretation of current HIV clinical practice guidelines (CPG).It will be included in the CHOICE counseling providing participants with patient-centered approach, specifically addresses the patient's expressed needs, problems, issues and concerns with a goal of providing accurate and unbiased information on available choices. After CHOICE counseling, if the participant chooses LAI-ART, the participant is referred to the SAVVY LAI-ART access team (SLAT) to facilitate access.
  Other Names: CHOICE counseling; HIV-ASSIST

SUMMARY:
Although there have been advances in antiretroviral treatment (ART) for HIV, adolescents and young adults living with HIV (AHIV) continue to have disparate HIV outcomes particularly viral suppression (VS), when compared to other populations likely related to multi-layered challenges (social determinants, cognitive development), system, and biomedical challenges including the reliance on oral ART as the only choice for HIV treatment. Given that approximately 1/3 of AHIV despite being in care fail to attain or sustain VS with resultant individual and public health risk, there is a need to develop real-world implementable interventions that can improve the participants virologic outcomes. The Strategies to AchieVe Viral Suppression for Youth with HIV (SAVVY) Study aims to 1) optimize personal ART choice by using the HIV-ASSIST clinical program to inform CHOICE counseling regarding an AHIV's preferred approach, including the possibility of long-acting injectable ART (LAI-ART); 2) facilitate access to the participants preferred choice through deploying a focused team to navigate barriers to attaining LAI-ART; and 3) decipher and address the patient, provider, and systemic barriers to the uptake and routinization of LAI-ART among AHIV by applying an implementation science framework and assessing cost-effectiveness providing critical data to support comprehensive approaches to optimizing ART and VS for AHIV, a key population identified in the Ending the HIV Epidemic in the United States Initiative.

DETAILED DESCRIPTION:
Adolescents and young adults (AHIV) ages 12-30 years have disproportionately poorer outcomes across the HIV care continuum, including lower rates of adherence to oral ART (oART) and viral suppression (VS) than older adults, correlating with individual risk of poor health and disease progression and public health risk of secondary transmission. AHIV are a priority population in the Ending the HIV Epidemic in the United States Initiative (EHE). Unique multi-layered factors (e.g., cognitive development, psychosocial determinants, system barriers) underlie AHIV's nonadherence and VS; therefore, AHIV-specific interventions are needed to address those factors and ultimately improve VS. Toward this aim, the investigators has shown that AHIV are more likely to be retained in care and achieve and maintain VS if cared for at clinics with youth-friendly structures and services, more likely to achieve VS with single tablet regimens (STR) vs. multi-tablet oral ART (oART) regimens, and have high interest in ART strategies not taken orally, specifically long-acting injectable ART (LAI-ART). These findings underscore the importance of engaging AHIV in decision-making and providing access to alternative biomedical strategies that obviate daily adherence, like LAI-ART, should the participant choose. Though uptake and roll-out has been slow, LAI-ART (cabotegravir/rilpivirine) administered q4-8 weeks has been approved for HIV treatment in those >12 years-old who have achieved VS-excluding up to 50% of all AHIV due to the decreased likelihood of VS. The investigators have reported provider biases and disparities in ART initiation by patient age and have concern that AHIV may have decreased access to LAI-ART, resulting in a tiered system that precludes LAI-ART access from those who may want and benefit from it most. AHIV need biomedical and care delivery innovations to address the challenges meeting EHE goals by optimizing feasibility of delivering novel biomedical tools for AHIV through minimizing medication and healthcare system barriers. The central hypothesis of the Strategies to AchieVe Viral Suppression for Youth with HIV (SAVVY) Study is that informed choice, counseling on ART options, and facilitating access, will increase rates of achieving and sustaining VS among AHIV. The study proposes to present and solicit informed choice of ART among both AHIV with and without VS, including facilitating LAI-ART (if VS can be achieved). For AHIV who prefer LAI-ART, the SAVVY intervention will support AHIV in successfully meeting or maintaining criteria (VL<50 copies/mL) for LAI-ART consideration, and deploy a focused team that facilitates access to LAI-ART. Study outcomes include VS and health-related quality of life (HRQOL) for AHIV undergoing the SAVVY intervention, identification of implementation barriers utilizing an established implementation science framework, and assessment of the cost-effectiveness of SAVVY using an economic-epidemiologic model. The investigators interdisciplinary team has expertise to implement the SAVVY study and the investigators anticipate that the results of The SAVVY study will inform the real-world implementation and optimization of LAI-ART AHIV toward reducing disparities in outcomes and ending the epidemic for the key population of AHIV.

ELIGIBILITY:
Inclusion Criteria:

* prescribed ART,
* willing to sign informed consent (including communication with one's primary HIV provider)

Exclusion Criteria:

* Relevant drug resistance mutations (per medical record) that compromises activity of Cabotegravir (CBG) + rilpivirine (RPV)
* disallowed medications,
* pregnancy.
* Mental health, cognitive, or behavioral dysfunction that in the opinion of the site PI would impair participation;
* severe illness/hospitalization at the time of enrollment,
* plan to move away in the next 12 months.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 288 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who reach viral suppression | 12 months
  Viral suppression (VL<20 copies/mL)

SECONDARY OUTCOMES:
Health related quality of life (HRQOL) as assessed by the Short Form 12 (SF-12) | 12 months
  Health related quality of life as measured by the SF-12. Score range: 0-100 with higher score indicating better quality of life.
Self-Efficacy as assessed by the Self-efficacy scale | 12 months
  Self-efficacy as measured by the self-efficacy scale. Scale range: 1 (cannot do it at all) to 10 (certain can do it).
Barriers to treatment adherence | 12 months
  Barriers to treatment as assessed by asking a series of 10 questions (Yes/No responses) addressing common Barriers to Treatment Adherence reported by individuals living with HIV, including housing, insurance, transportation, and other domains. Score range: 0-10 with a higher number of items reported equating to greater number of barriers.
HIV stigma scale | 12 months
  HIV stigma as measured by the HIV stigma scale. The questionnaire uses a 4-point Likert scale ranging from strongly disagree (1) to strongly agree (4). Possible score range of 3 to 12; higher scores reflect a higher level of perceived HIV-related stigma.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Agwu, MD, SCM, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No